CLINICAL TRIAL: NCT03939819
Title: Comparison Between Endoscopic vs. Suction Calibration System on Number of Staple Load Firings, Operative Duration, Cost, and Gastro-esophageal Reflux Disease Following Laparoscopic Sleeve Gastrectomy: is There a Difference
Brief Title: Endoscopic vs. Suction Device Calibration in Sleeve Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Elizabeth Hechenbleikner, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00108907
Record Dates: First submitted 2019-05-03; First posted 2019-05-07 (Actual); Results first posted 2023-03-07 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Gastrectomy; Obesity
Keywords: weight loss surgery; laparoscopic sleeve gastrectomy; suction calibration system; bariatric surgery
MeSH Terms: conditions — Obesity | interventions — Endoscopy, Digestive System; Calibration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- ViSiGi® 3D suction calibration device (Experimental): The ViSiGi® 3D is the first calibration system specifically intended for use during sleeve gastrectomy.ViSiGi 3D®is a non-sterile, single patient use device. The device comprises a tube with a closed, rounded tip, and holes at the distal end. The proximal end of ViSiGi 3D® includes an integral suction regulator and vented On/Off valve.
  Advantages of ViSiGi® 3D device include simplification of sleeve calibration in addition to suctioning the stomach and performing leak tests all with one device making operative steps simpler for both the anesthesiology team and surgeons. Since it is single patient use it does not require reprocessing.
  Interventions: Device: ViSiGi® 3D suction calibration device
- Esophagogastroduodenoscopy (EGD) calibration (Active Comparator): Gastroscope, similar to The ViSiGi device, have suction, calibration, and leak testing capabilities.
  Interventions: Device: Esophagogastroduodenoscopy (EGD) calibration

INTERVENTIONS:
Device: ViSiGi® 3D suction calibration device — ViSiGi 3D®is a non-sterile, single patient use device. The device comprises a tube with a closed, rounded tip, and holes at the distal end. The proximal end of ViSiGi 3D® includes an integral suction regulator and vented On/Off valve.
  Arms: ViSiGi® 3D suction calibration device
Device: Esophagogastroduodenoscopy (EGD) calibration — Gastroscope is an illuminated optical, slender and tubular instrument (a type of borescope) used in esophagogastroduodenoscopy.
  Arms: Esophagogastroduodenoscopy (EGD) calibration

SUMMARY:
This study aims to compare the difference in staple usage and post-operative GERD (heartburn) between patients that had an endoscope used versus patients that had a suction calibration system used on them during "laparoscopic sleeve gastrectomy" (LSG).

DETAILED DESCRIPTION:
There are multiple choices for a surgeon and their patient when it comes to weight loss surgery. One of those options is a procedure called a "laparoscopic sleeve gastrectomy" (LSG). In this procedure the majority of the patient's stomach is removed leaving behind a stapled "sleeve" about the same size as the patient's esophagus.

During this procedure there are three main devices that surgeon inserts through the mouth and in to the stomach to calibrate the size of the "sleeve". They can use a standard weighted bougie, an endoscope, or a suction calibration device. This study aims to compare the difference in staple usage and post-operative GERD (heartburn) between patients that had an endoscope used versus patients that had a suction calibration system used on them during LSG.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* agreed with a surgeon that laparoscopic sleeve gastrectomy (LSG) is the best choice

Exclusion Criteria:

* Had prior gastric surgery or bariatric surgery (including prior adjustable gastric band and/or sleeve gastrectomy)
* Concomitant hiatal surgery
* Paraesophageal hernia at time of surgery
* Any subject with prescribed immunosuppressive drugs.
* In the opinion of investigator, subject is not eligible to participate in the study.
* If patient is a female and becomes pregnant at any time during the study duration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Hechenbleikner, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital Midtown, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
The study team does not plan to make the data available to other researchers.

RESULTS

PARTICIPANT FLOW:
Groups:
- ViSiGi® 3D Suction Calibration Device: The ViSiGi® 3D is the first calibration system specifically intended for use during sleeve gastrectomy.ViSiGi 3D®is a non-sterile, single patient use device. The device comprises a tube with a closed, rounded tip, and holes at the distal end. The proximal end of ViSiGi 3D® includes an integral suction regulator and vented On/Off valve.
  Advantages of ViSiGi® 3D device include simplification of sleeve calibration in addition to suctioning the stomach and performing leak tests all with one device making operative steps simpler for both the anesthesiology team and surgeons. Since it is single patient use it does not require reprocessing.
  ViSiGi® 3D suction calibration device: ViSiGi 3D®is a non-sterile, single patient use device. The device comprises a tube with a closed, rounded tip, and holes at the distal end. The proximal end of ViSiGi 3D® includes an integral suction regulator and vented On/Off valve.
Period: Overall Study
Arm/Group | ViSiGi® 3D Suction Calibration Device | Esophagogastroduodenoscopy (EGD) Calibration
Started | 50 | 56
Completed | 48 | 56
Not Completed | 2 | 0
Not completed — Death | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ViSiGi® 3D Suction Calibration Device | Esophagogastroduodenoscopy (EGD) Calibration | Total
Number analyzed (Participants) | 50 | 56 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.80 (11.14) | 43.90 (12.13) | 43.38 (11.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 47 | 89
  Male | 8 | 9 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 40 | 47 | 87
  Unknown or Not Reported | 9 | 9 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 34 | 39 | 73
  White | 13 | 15 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 50 | 56 | 106
Mean total body weight at 1-2 months prior to surgery [Mean (Standard Deviation); unit: Kg] — Population: Number analyzed in row differs from overall because there was one pre-op weight missing in each group.
  Kg
    number analyzed (Participants) | 49 | 55 | 104
    (all) | 138.1 (28.7) | 135.7 (27.8) | 137.0 (29.4)

OUTCOME MEASURES:

1. Primary Outcome: Number of Staple Load Firings
Description: Staple usage will be recorded during the weight loss surgery procedure.
Time Frame: During sleeve gastrectomy (up to 5 hours)
Measure: Mean (Standard Deviation); unit: Number of staples
Arm/Group | ViSiGi® 3D Suction Calibration Device | Esophagogastroduodenoscopy (EGD) Calibration
Number analyzed (Participants) | 50 | 56
Number of staples | 5.26 (0.78) | 5.42 (0.89)

2. Secondary Outcome: Operative Duration (Time)
Description: Surgery start and completion time will be recorded, and operative duration will be calculated
Time Frame: During sleeve gastrectomy (up to 5 hours)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | ViSiGi® 3D Suction Calibration Device | Esophagogastroduodenoscopy (EGD) Calibration
Number analyzed (Participants) | 50 | 56
minutes | 93.38 (28.10) | 94.42 (36.50)

3. Secondary Outcome: Intra-operative Cost for Patients
Description: Cost data (administrative data) will be retrieved from internal database
Time Frame: During sleeve gastrectomy (up to 5 hours)
Population: Data for this study outcome was not collected due to internal limitations of the study.
Arm/Group | ViSiGi® 3D Suction Calibration Device | Esophagogastroduodenoscopy (EGD) Calibration
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: GERD Symptom Severity Score
Description: GERD-HRQL questionnaire will be administered pre-operatively and post-operatively. The instrument contains a total of 10 scaled items which are scored, and a patient-reported global satisfaction assessment which is not added to the total GERD-HRQL score. Higher score correlates with worse outcome. Scale: No symptoms = 0; Symptoms noticeable, but not bothersome = 1; Symptoms noticeable and bothersome, but not every day = 2; Symptoms bothersome every day = 3; Symptoms affect daily activities = 4; Symptoms are incapacitating, unable to do daily activities = 5
Time Frame: 1-2 months prior to surgery, 3 weeks post-operatively (+/- 2 weeks), 12 months post-operatively (+/- 12 - 24 months)
Population: Number of participants analyzed only included patients that were able to complete the questionnaire at each time point, which is different for each follow up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ViSiGi® 3D Suction Calibration Device | Esophagogastroduodenoscopy (EGD) Calibration
Number analyzed (Participants) | 50 | 56
score on a scale
  GERD-HRQL Score at 1-2 months prior to surgery | 4.54 (5.7) | 3.82 (5.67)
  GERD-HRQL Score at 3 weeks post-operatively (+/- 2 weeks): number analyzed (Participants) | 35 | 32
  GERD-HRQL Score at 3 weeks post-operatively (+/- 2 weeks) | 3.00 (4.33) | 5.66 (9.56)
  GERD-HRQL Score at 12 months post-operatively (+/- 12 - 24 months): number analyzed (Participants) | 43 | 41
  GERD-HRQL Score at 12 months post-operatively (+/- 12 - 24 months) | 2.58 (4.15) | 2.64 (3.79)

5. Secondary Outcome: Body Weight
Description: Total body weight was calculated in Kg.
Time Frame: 3 weeks post-operatively (+/- 2 weeks), 12 months post-operatively (+/- 12 - 24 months)
Population: Unable to get reliable weight loss data for the early post-op time frame for 3 weeks post-operatively (+/- 2 weeks).
  Number of participants analyzed for the long-term follow up included patients that completed the appointment including weight check.
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | ViSiGi® 3D Suction Calibration Device | Esophagogastroduodenoscopy (EGD) Calibration
Number analyzed (Participants) | 31 | 38
Kg
  Body weight at 3 weeks post-operatively (+/- 2 weeks): number analyzed (Participants) | 0 | 0
  Body weight at 12 months post-operatively (+/- 12 - 24 months) | 108.2 (24.9) | 106.7 (24.5)

ADVERSE EVENTS:
Time Frame: From date of surgery up to 12 months post-operatively (+/- 12 - 24 months).
Description: The PI will be informed of serious adverse events (AEs) as soon as they occur by Co-Investigators (i.e.,surgeons performing sleeve gastrectomy) and/or the study coordinator and notify the Medical board (MB) within 48 hours of becoming aware of the event. The PI will report serious AEs and unanticipated problems (UPs) to his or her IRB within 5 business days of becoming aware of the event. Data collection for Adverse events is still ongoing.
Arm/Group | ViSiGi® 3D Suction Calibration Device | Esophagogastroduodenoscopy (EGD) Calibration
All-Cause Mortality (participants affected / at risk) | 2/50 | 0/56
Serious Adverse Events (participants affected / at risk) | 2/50 | 0/56
Other Adverse Events (participants affected / at risk) | 0/50 | 0/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ViSiGi® 3D Suction Calibration Device (N=50) | Esophagogastroduodenoscopy (EGD) Calibration (N=56)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cerebral Accident (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-17): https://cdn.clinicaltrials.gov/large-docs/19/NCT03939819/Prot_SAP_000.pdf